CLINICAL TRIAL: NCT03259048
Title: Role of Ultrasound in Diagnosis of Acute Abdomen in Pediatric Group
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohmed abdelwahab, Resident of Radiology Department - Assiut University, Assiut University
Other Study IDs: Assiut University Hospitals
Record Dates: First submitted 2017-08-19; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Ultra Sound in Diagnosis of Acute Abdomen in Pediatric Group

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric group: pediatric group from age of one day to eighteen years.
  Interventions: Diagnostic Test: Abdominal ultrasound

INTERVENTIONS:
Diagnostic Test: Abdominal ultrasound — Abdominal ultrasound will be used in the diagnosis of acute abdomen in pediatric group.

SUMMARY:
Acute abdomen can be defined as "A syndrome induced by wide variety of pathological conditions that require emergent medical or more often surgical management" [1].There are a plethora of causes that can lead to acute abdomen in children, they vary depending on the ages of the children and can be divided into diseases that can be treated with medical care and those in which emergency surgical intervention must be considered [2]. Ultrasonography is the initial choice in the diagnosis of the different causes of acute abdomen in children [3, 4]. It is very useful as it is non-invasive, cost- effective, repetitive, with no radiation exposure, as good as laparoscopy, can be done even in patients with scarred abdomen [5].

DETAILED DESCRIPTION:
-Patient preparation:

* No specific preparation is needed.
* Demographic data including age, sex, detailed history, clinical presentation, laboratory tests, and data of any other investigations or operation will be obtained.
* Clinical examination will be done in emergency pediatric unit for provisional diagnosis.

  -Study instruments:• Patients will examined by Grey-Scale Ultrasonography (U/S) combined with Color Doppler Ultrasonography (CDUS).

  3-Technique of examination
* will be in supine position.
* Patient First examination of whole abdomen will be done by Grey -Scale U/S using both 3.5 MHZ and 7.5 MHZ transducers .It will be done in both longitudinal ( parallel to long axis of the patient ) and transverse ( perpendicular to long axis of the patient ) orientation .
* Then finally examination by Color Doppler US will be done for assessment of organ perfusion and diagnosing inflammation.

ELIGIBILITY:
Inclusion Criteria:

* -In this study, 100 patients referred from the emergency Pediatric Unit for the assessment of the cause of acute abdomen.

Exclusion Criteria:

* - Patients of age group above 18 years
* Patients with trauma.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients referred from the emergency Pediatric Unit for the assessment of the cause of acute abdomen from age of 1 day to 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of ultrasound in diagnosis of acute abdomen | 2 years
  efficacy of ultrasound in diagnosis of acute abdomen

IPD SHARING:
Plan to Share IPD: No